CLINICAL TRIAL: NCT04002336
Title: Testing a Smart Phone App to Enhance Voice Therapy Adherence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vrushali Angadi (Other)
Responsible Party: Sponsor-Investigator, Vrushali Angadi, Assistant Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 44183
Record Dates: First submitted 2019-06-26; First posted 2019-06-28 (Actual); Last update posted 2019-06-28 (Actual); Status verified 2019-06

CONDITIONS: Voice Disorders
Keywords: adherence
MeSH Terms: conditions — Voice Disorders

STUDY DESIGN:
Who Masked: Participant
Masking Description: Single-blinded to primary outcome measure
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional Voice Therapy (Active Comparator): Standard of care (traditional) voice therapy.
  Interventions: Behavioral: Traditional Voice therapy
- App Group (Experimental): Voice therapy using a smartphone app.
  Interventions: Behavioral: Voice Therapy App

INTERVENTIONS:
Behavioral: Traditional Voice therapy — Traditional method of voice therapy
  Other Names: Vocal Function Exercises
  Arms: Traditional Voice Therapy
Behavioral: Voice Therapy App — Smartphone app, which allows participants to record home practice sessions in real time and upload sessions to the app server for the clinician to access and track.
  Other Names: Vocal Function Exercises
  Arms: App Group

SUMMARY:
The current project is designed as phase 1 study conducted to improve/enhance normal voice. Fifteen Thirty non-treatment seeking individuals, with no identifiable vocal pathology on laryngeal examination, will be randomized to one of two groups; 1) Voice therapy delivery without App (control/standard of care), 2) Voice therapy delivery with app (experimental). Participants in both groups will attend weekly voice therapy sessions (for 6 weeks) with the PI and Co- I (Joseph Stemple). Control group participants will be provided with an audio file of the exercises, and an exercise log sheet to track progress. Experimental group participants will use the smartphone app, which allows participants to record home practice sessions in real time and upload sessions to the app server for the clinician to access and track. Three-wave surveys will be conducted at the baseline, four weeks and 6 weeks after the intervention. Other data sources include study administration, exercise logs, app data, and clinical assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Adults > 18 years
2. Non-smokers
3. Hearing level within normal limits
4. Absence of vocal fold pathology as confirmed by MD on laryngeal examination
5. Agree to avoid vocally abusive behaviors for the entirety of the study

Exclusion Criteria:

1. Apple phone (iOS)
2. Impaired hearing
3. Uncontrolled asthma
4. Smoking
5. H/o vocal fold surgery
6. Presence of vocal fold pathology
7. Previous history of experience with VFE performance
8. Non-English speaking participants

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
Adherence | 6 weeks
  Number of completed home practice sessions

SECONDARY OUTCOMES:
MPT (maximum phonation time) | 6 weeks
  Maximum phonation time

CONTACTS AND LOCATIONS:
Overall Officials: Vrushali Angadi, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No